CLINICAL TRIAL: NCT01496482
Title: Comparison of Evaporimetry With the Established Methods of Tear Film Measurement
Status: Completed | Type: Observational
Sponsor: University of Zagreb (Other)
Responsible Party: Principal Investigator, Igor Petricek, Ophthalmologist, MD, PhD, Head of the Ocular Electrophysiology and Ultrasound Laboratory, University of Zagreb
Other Study IDs: UZagreb Eye 1; Dry Eye 1 (Other: Zagreb University Hospital Eye Department, Zagreb, Croatia)
Record Dates: First submitted 2011-12-03; First posted 2011-12-21 (Estimated); Last update posted 2011-12-22 (Estimated); Status verified 2011-12

CONDITIONS: Dry Eye Syndromes
Keywords: Dry eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients without dry eye symptoms: Patients without dry eye symptoms as measured by standard questionnaire.
  Interventions: Other: Only measurements done on subjects in both groups.
- Patients with dry eye symptoms: Patients with dry eye symptoms as measured by standard questionnaire.
  Interventions: Other: Only measurements done on subjects in both groups.

INTERVENTIONS:
Other: Only measurements done on subjects in both groups. — As study compared specific diagnostic procedures, no intervention was done or compared.

SUMMARY:
Purpose:

To establish whether there is a correlation between dry eye symptoms, age and gender, a difference in symptom intensity in different times of the day, which test (Schirmer or TBUT) better correlates with dry eye symptoms, whether it is possible to reliably use cheap, easy to use hygrometer in everyday clinical setting, and finally whether there is statistically significant correlation between applied tests (TBUT, Schirmer and evaporimetry).

Methods:

Subjects: 45 in group without dry eye related symptoms, and 45 in group with symptoms.

Examination included structured case history (questionnaire), slit lamp examination with fluorescein staining, periocular evaporimetry, TBUT test and Schirmer test.

DETAILED DESCRIPTION:
Purpose:

The purpose of this study was to establish whether there is a correlation between dry eye symptoms, age and gender, any difference in symptom intensity in different times of the day, which test (Schirmer or TBUT) better correlates with dry eye symptoms, whether it is possible to reliably use cheap, easy to use hygrometer in everyday clinical setting, and, finally, whether there is statistically significant correlation between applied tests (TBUT, Schirmer and evaporimetry).

Methods:

Subjects were divided in two groups: 45 in group without dry eye related symptoms, and 45 in group with symptoms.

Examination was performed in the following sequence:

1. structured case history (questionnaire),
2. evaporimetry
3. slit lamp examination with fluorescein staining,
4. TBUT test and
5. Schirmer test I (without anesthetic, closed eyes)

Case history consisted of the following questions:irritation more pronounced on wind? irritation during reading and/or watching TV or computer? irritation more pronounced during winter? gritty sensation in the eyes? irritation more pronounced in the morning or evening? All answers, except to the last question, were graded from 0 (no complaints) to 3 (severe).

Evaporimetry was performed using commercially available hygrometer from HYGROTEC (Titisee-Neustadt, Germany), installed in swimming goggles with its front part sawn off.

First measurement was performed by measuring for 5 minutes with eyes closed. Second measurement also lasted 5 minutes, with eyes kept open, normal blinking, and with subject fixating at one point in distance, with no eye movements.

Measured parameters included:

basal φ (%): relative environment humidity before measurement basal T: environment temperature before measurement closed eye φ (%): relative humidity in front of closed eye open eye φ (%): relative humidity in front of open eye C/O: ratio of φ (%) closed/open eye

ELIGIBILITY:
Inclusion Criteria:

* patients with or without dry eye symptoms

Exclusion Criteria:

* minors
* pregnant women
* patients with acute eye conditions (inflammation, allergy, trauma)
* patients with chronic eye diseases requiring continuous topical treatment (i.e.glaucoma)
* ocular surface scarring
* patients who did not sign informed consent.

Ages: 18 Years to 61 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients were volunteers who came for a standard ophthalmological exam in Zagreb University Hospital Eye Clinic, and whose enrollment was based on convenience sampling.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2008-09; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Tear evaporation | 10 minutes
  Five minutes of tear evaporation measurement with eyes closed and five with open, normal blinking.

SECONDARY OUTCOMES:
Comparison of tear evaporation to symptoms score | 15 minutes (10 minutes tear evaporation, 5 minutes symptoms score recording)
  Tear evaporation measurement compared to dry eye symptoms score (0-15 points).
Comparison of tear evaporation to Tear Film Break-up Time (TBUT) | 15 minutes (10 minutes evaporation measurement, 5 minutes TBUT measurement)
  Comparison of tear evaporation to Tear Film Break-up Time (seconds).
Comparison of tear evaporation to Schirmer test | 15 minutes (10 minutes tear evaporation measurement, 5 minutes Schirmer test)
  Comparison of tear evaporation to Schirmer test (mm)
Comparison of tear evaporation to corneal staining | 12 minutes (10 minutes tear evaporation measurements, 2 minutes corneal staining assessment)
  Comparison of tear evaporation to corneal staining using fluorescein (score 1-3):
  1:5-10 corneal stains at six o'clock; 2: 10-25 corneal stains; 3: more than 26 diffuse corneal stains
Comparison of tear evaporation to conjunctival hyperemia | 11 minutes (10 minutes evaporation measurement, 1 minute conjunctival hyperemia assessment)
  Comparison of tear evaporation to conjunctival hyperemia (score 1-3):
  1: minimal; 2: moderate; 3: severe

CONTACTS AND LOCATIONS:
Overall Officials: Igor Petricek, MD, PhD, Principal Investigator — Zagreb University Hospital Eye Department, Zagreb, Croatia
Locations (1):
- Zagreb University Hospital Eye Department, Zagreb, Croatia